CLINICAL TRIAL: NCT01171027
Title: Prospective Multicenter Human Randomized Controlled Evaluation of NOTES® Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Natural Orifice Surgery Consortium for Assessment and Research (Other)
Collaborators: American Society for Gastrointestinal Endoscopy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NOTES® Trial
Record Dates: First submitted 2010-07-26; First posted 2010-07-28 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-11

CONDITIONS: Gall Bladder Diseases
Keywords: Cholecystectomy; NOTES; Transvaginal; Transgastric; Natural orifice; Gallbladder removal
MeSH Terms: conditions — Gallbladder Diseases | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NOTES(R) Cholecystectomy (Experimental): Natural Orifice Translumenal Endoscopic Surgery techniques
  Interventions: Procedure: NOTES Cholecystectomy
- Laparoscopic Cholecystectomy (Active Comparator): Laparoscopic Cholecystectomy
  Interventions: Procedure: NOTES Cholecystectomy; Procedure: Laparoscopic Cholecystectomy

INTERVENTIONS:
Procedure: NOTES Cholecystectomy — The transvaginal NOTES approach is accomplished by performing a posterior colpotomy. Instead of a conventional laparoscope, a flexible endoscope is used in order to provide working channels and visualization. The gallbladder is removed through the vaginal incision. The transgastric cholecystectomy requires the flexible endoscope to be placed orally. A gastrotomy is made through the stomach wall allowing the flexible endoscope to pass into the abdominal cavity. The gallbladder is removed from the abdominal cavity into the stomach and ultimately out the mouth. The goal of NOTES is to develop further so either of these approaches will not require any incisions in the abdominal wall.
Procedure: Laparoscopic Cholecystectomy — This technique utilizes the introduction of a laparoscope through a 1 cm incision in the fascia in or around umbilicus. Usually three additional 0.5- 1.0 cm incisions are employed for surgical instrumentation. Once separated from its attachments, the gallbladder is usually removed through the umbilical port. Sutures are used to close the larger port sites. The most devastating complication is injury to the major bile ducts which is avoided to the extent possible (incidence .2 to less than .01%)5 by careful visualization of the ductal structures.
  Arms: Laparoscopic Cholecystectomy

SUMMARY:
This study is designed to be a United States multicenter prospective randomized controlled non-inferiority evaluation of transgastric and transvaginal Natural Orifice Translumenal Endoscopic Surgery (NOTES) cholecystectomy compared to laparoscopic cholecystectomy in elective surgery patients. Up to 200 patients will be enrolled to obtain 70 NOTES cholecystectomies (35 transgastric and 35 transvaginal) and 70 laparoscopic cholecystectomies on a randomized basis. In order to evaluate the hypothesis that NOTES cholecystectomy has equivalent safety and efficacy to laparoscopic cholecystectomy, clinical and administrative outcomes will be measured.

DETAILED DESCRIPTION:
Primary To assess the safety and efficacy of transgastric and transvaginal cholecystectomy compared to conventional laparoscopic cholecystectomy.

To assess pain associated with transgastric and transvaginal cholecystectomy compared to conventional laparoscopic cholecystectomy.

Secondary To assess cosmesis associated with transgastric and transvaginal cholecystectomy compared to conventional laparoscopic cholecystectomy.

To assess objective operative cost and logistical comparisons between transgastric and transvaginal cholecystectomy compared to conventional laparoscopic cholecystectomy.

To identify unforeseen barriers to transgastric or transvaginal surgery adoption.

ELIGIBILITY:
Inclusion Criteria:

* Competent male or female subjects, between the ages of 18-75 and who present for elective cholecystectomy will be offered participation in this study.
* Male subjects must be willing to have the cholecystectomy by either the laparoscopic or transgastric NOTES approach.
* Female subjects must be willing to have the cholecystectomy by either the laparoscopic or either the NOTES approaches (transgastric and/or transvaginal) being performed at the site.
* Patients offered participation in this study must provide written, informed consent and meet the following criteria prior to randomization.
* Diagnosis of benign gallstone disease which requires cholecystectomy.
* ASA Class 1 or 2.
* Willingness to have laparoscopic cholecystectomy performed and have research data collected for control group.
* Willingness to have abdomen photographed (for cosmesis assessment).
* For sites performing transgastric NOTES approach

  * Willingness to have cholecystectomy performed via NOTES transgastric approach.
  * Willingness to have NOTES procedure videotaped.
* For sites performing transvaginal NOTES approach - Female subjects only

  * Willingness to have cholecystectomy performed via NOTES transvaginal approach.
  * Willingness to have intra-abdominal procedure digitally recorded.
  * Pelvic examination in the past 12 months without significant pathology.

Exclusion Criteria:

* Pregnant women.
* Obese patients (BMI > 35).
* Patients with severe medical comorbidities (ie, NOT ASA Class 1 or 2) will be excluded such as:
* Chronic renal failure
* Chronic liver disease
* Congestive heart failure
* Patients with a presumed gallbladder malignancy.
* Patients with a history of prior open abdominal or laparoscopic or transvaginal surgery. However patients with prior appendectomy, tubal ligation or Cesarean section will be included.
* Patients who are taking immunosuppressive medications and/or immunocompromised.
* Patients with a prior history of perineal trauma leading to significant alteration of vaginal anatomy.
* Patients with a history of ectopic pregnancy, pelvic inflammatory disease, large fibroids or severe endometriosis.
* Patients with known common bile duct stones. (ie, not cleared prior to surgery). Patients with common bile duct stones discovered intra-operatively will remain in the study.
* Patients on anticoagulation drugs other than once daily aspirin. Abnormal blood coagulation tests. Minimal abnormalities may be allowed at the discretion of site principal investigator.
* Gallstones> 2.5cm in diameter.
* Presence of untreated esophageal stricture.
* Surgically altered gastric anatomy or severe uncorrected paraesophageal types 2, 3 or 4.
* Unwillingness to consent to NOTES procedure(s).
* Acute cholecystitis or cholangitis
* For sites performing transgastric NOTES approach

  * Contraindicated for esophagogastroduodenoscopy (EGD).
  * Patients with hypersecretory states.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-06 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and efficacy of transgastric and transvaginal cholecystectomy compared to conventional laparoscopic cholecystectomy. | 4 weeks post surgery

SECONDARY OUTCOMES:
To assess pain associated with transgastric and transvaginal cholecystectomy compared to conventional laparoscopic cholecystectomy. | 4 weeks post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Steven Schwaitzberg, MD, Principal Investigator — Cambridge Health Alliance; Michael L. Kochman, MD, Principal Investigator — University of Pennsylvania
Locations (6):
- United States (6):
  - University of California at San Diego, San Diego, California
  - Yale University, New Haven, Connecticut
  - Northwestern University, Chicago, Illinois
  - Baystate Medical Center, Springfield, Massachusetts
  - Ohio State University, Columbus, Ohio
  - Oregon Clinic, Portland, Oregon

REFERENCES:
- See also: NOSCAR web site — http://www.noscar.org